CLINICAL TRIAL: NCT02819193
Title: Using Mother's Raw Milk Could Improve Breastfeeding in Hospitalized Neonates
Acronym: DOAL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0379
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Breastfeeding
Keywords: Breastfeeding; mother's milk; breast milk; raw milk; neonate; Neonatal intensive care unit (NICU)
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- exposed group : early raw mother's own milk: The use of raw MOM is considered as "early" when it begins before day 7.
  Interventions: Other: raw mother's own milk
- unexposed group : no use of raw mother's own milk: Neonates who receive, or not, raw MOM before day 7.

INTERVENTIONS:
Other: raw mother's own milk — Infants receive mother's own milk before day 7.
  Groups: exposed group : early raw mother's own milk

SUMMARY:
Despite the importance of breast milk for sick or preterm neonates, there is currently no consensus regarding the use of raw mother's own milk (MOM) in neonatal units. The aims of this study are to: (a) describe factors associated with the use of raw MOM; (b) investigate the association between early use of raw MOM and breastfeeding continuation at discharge and up to 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Admitted neonates between April 2012 and June 2013 are eligible if they are intended to be breastfeed and hospitalized ≥7 days

Exclusion Criteria:

- Neonates with parents not fluent in French.

Max Age: 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates from two French participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Maternal breastfeeding | up to 6 months
  Maternal breastfeeding is defined as the consumption of any MOM. It is classed as "exclusive" when all the fed milk will be MOM or "partial" when it will be completed by other milk or food.

CONTACTS AND LOCATIONS:
Overall Officials: Céline Fischer Fumeaux, MD, Principal Investigator — Service de Réanimation Néonatale et Néonatologie, Hôpital Femme Mère Enfant, Bron, France
Locations (1):
- Service de Réanimation Néonatale et Néonatologie, Hôpital Femme Mère Enfant, 32 Avenue Doyen Jean Lépine, Bron, France